CLINICAL TRIAL: NCT00831480
Title: Neoadjuvant Everolimus (RAD001)for Advanced RCC Before Cytoreductive Nephrectomy, With Correlative Tumor Studies (Protocol #: 06-08-20-01)
Brief Title: Everolimus (RAD001) For Advanced Renal Cell Carcinoma (RCC) Before Kidney Removal
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in accrual and by the order of the cancer center.
Sponsor: Linda C. Higgins (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor-Investigator, Linda C. Higgins, Study Contact, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-23409
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2014-12

CONDITIONS: Kidney Cancer
Keywords: Renal cell carcinoma; Everolimus; Neoadjuvant; advanced kidney cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All subjects will take everolimus
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — everolimus 10 mg PO once daily for 3-5 weeks followed by removal of the kidney. Everolimus will begin again between 2 to 4 weeks after surgery.
  Other Names: RAD001; Afinitor

SUMMARY:
The purpose of this multicenter, pilot, open-label, Phase II clinical trial is to discover if Everolimus(RAD001) is safe and effective in people who have advanced kidney cancer (renal cell carcinoma - RCC).

Since 2002, Everolimus has been studied in more than 2500 patients with various types of cancer as a single agent (a drug that is used alone to treat the cancer) or in combination with a number of well known anticancer therapies. Various studies, in animals such as in mice with cancer and in humans with cancer have shown that Everolimus can slow the growth of cancer.

Everolimus will be taken in pill form by mouth daily for 3-5 weeks followed by surgery to remove the effected kidney. After 2-4 weeks following the surgery, Everolimus will be resumed at the same dose.

DETAILED DESCRIPTION:
Everolimus has significantly improved outcomes following prior therapy. This study is a biomarker driven Phase II trial that will assess the activity of everolimus as first-line therapy for renal cell carcinoma. Following initial kidney tumor biopsy, everolimus is administered for 3-5 weeks before cytoreductive nephrectomy and everolimus is then resumed and continued until tumor progression or intolerable toxicities. Any correlation of tumor tissue biomarker changes from initial biopsy to nephrectomy specimen with long-term progression-free survival will be determined. This trial may enable the identification of factors predictive of significant benefit from everolimus administered as first-line therapy by employing the neoadjuvant therapy paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Advanced (metastatic) RCC
* Histology: clear cell, papillary or chromophobe
* 3 out 6 risk factors (by Memorial Sloan Kettering Cancer Center criteria and one additional criterion: multiple sites of metastasis) or not candidates for or refuse sunitinib.
* Must have at least one measurable metastatic site according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria that has not been previously irradiated.
* Must be deemed surgical candidates for cytoreductive nephrectomy by the urologist.
* Age 18 years of age or older
* Eastern Cooperative Oncology Group (EGOG) PS 0-2
* Adequate bone marrow function
* Adequate liver function as shown by:
* Adequate renal function
* Fasting serum cholesterol AND fasting triglycerides within normal limits
* Signed informed consent

Exclusion Criteria:

* Collecting duct, medullary histologies or sarcomatoid differentiation.
* Central Nervous System (CNS) or leptomeningeal metastases.
* Inappropriate candidates for cytoreductive nephrectomy or who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* severely impaired lung function
* uncontrolled diabetes
* active (acute or chronic) or uncontrolled severe infections
* liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Ineligible for cytoreductive nephrectomy
* Current or prior systemic anticancer therapies (including chemotherapy, antibody based therapy, or investigational drugs)
* Other malignancies within the past 3 years except for localized carcinoma of the cervix, basal or squamous cell carcinomas of the skin, or localized prostate cancer with Gleason Score less than 7 treated with radiation or surgery and no evidence of progression.
* Major surgery (defined as requiring general anesthesia) or significant traumatic injury within 4 weeks of start of enrollment
* Anticipated major surgery (other than CN) during the course of the study
* A known history of HIV seropositivity
* Hepatitis C seropositivity
* Chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Immunization with attenuated live vaccines within one week of study entry or during study period
* Known hypersensitivity to RAD001 (everolimus) or other rapamycins or to its excipients
* Impairment of gastrointestinal function or gastrointestinal disease
* Active, bleeding diathesis
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
* History of noncompliance to medical regimens
* Unwilling to or unable to comply with the protocol including mandated biopsies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-04; Primary Completion 2013-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilad E. Amiel, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifteen subjects signed informed consents. Out of that 15, 9 took at least one dose of study drug.
Groups:
- Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore: All subjects will take everolimus
  everolimus: everolimus 10 mg PO once daily for 3-5 weeks followed by removal of the kidney. Everolimus will begin again between 2 to 4 weeks after surgery.
Period: Overall Study
Arm/Group | Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore
Started | 9
Completed | 7
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Patients with clinically measurable metastatic RCC
Arm/Group | Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 58.9 [46 to 70]
Age, Categorical [Count of Participants; unit: Participants] — Image and biopsy proven metastatic RCC
  Participants
    <=18 years | 0
    Between 18 and 65 years | 7
    >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Evidence of Metastatic Disease [Number; unit: participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Disease Progression Diagnosed by Biopsy
Description: Clinical progression validated by biopsy of metastatic site. Progression-free survival (PFS) will be measured from the post-op treatment start date to either the date the patient is first recorded as having disease progression, or the date of death if the patient dies due to any causes before progression. If a patient is lost to follow-up or removed for toxicities, the patient will be censored as of the last date of contact. Patients who start a new treatment before they progress will be censored as of the date of start of the new treatment. If a patient has not progressed or died, PFS is censored at the date of last follow-up. Patients removed from therapy with everolimus due to toxicities will not be included in the PFS estimation.
Time Frame: up to one year
Measure: Number; unit: participants
Arm/Group | Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore
Number analyzed (Participants) | 9
participants | 9

ADVERSE EVENTS:
Arm/Group | Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore (N=9)
Kidney Injury (Surgical and medical procedures) | 1 (1) — 6 days after operation, creatinine rose.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Everolimus "RAD001" for Advanced RCC Before Cytore (N=9)
mucositis of tongue (Skin and subcutaneous tissue disorders) | 6 (6) — mucositis of tongue

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No